CLINICAL TRIAL: NCT05877794
Title: Does the Central Venous Puncture Needle Need to be 7 cm? ; Safety and Usefulness of Needle Length Adjustment Method Using Suture Wing
Brief Title: Does the Central Venous Puncture Needle Need to be 7 cm?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, associate professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AJIRB-MED-INT-22-188
Record Dates: First submitted 2022-06-17; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Central Venous Catheters

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- wing group (Experimental)
  Interventions: Device: central venous catheter insertion

INTERVENTIONS:
Device: central venous catheter insertion — All patients were under trendlenburg position (10 degrees) and disinfected for CVC catheterization. After attaching 2 suture wings of 18G single catheter set to the insertion needle in the 7 Fr or 8 Fr central catheter set, check the IJV to be punctured with an ultrasonic probe. The IJV is punctured using a cross sectional image confirmed at the cricoid cartilage level. After confirming the needle tip on the ultrasound image and blood coming out, the guide wire is mounted on the IJV and then a CVC catheter (arrow international INC) ., USA) is inserted. All actions are performed by a specialist who has more than 30 CVC catheterization experiences using ultrasound, and the occurrence of side effects and the time from puncture to guide wire entry are recorded by another researcher. After the procedure, the researcher who directly performed the procedure records the difficulty or difference compared to when using a conventional needle that does not have a suture wing installed.

SUMMARY:
The central venous catheter (CVC) has been used for the first time in clinical use in 1921 and has been used worldwide by 2023. Although there are differences between studies, it is reported that side effects occur in approximately 5-20% of patients undergoing CVC. Common side effects include hematoma, venous puncture, arterial puncture, and pneumothorax, and horner syndrome is also reported in 5% of cases. In particular, in the case of the internal jugular vein (IJV), the possibility of puncture of the internal carotid artery is higher than that of other sites, and the puncture level also varies depending on the depth of needle insertion, which in some cases can cause very serious side effects. The incidence rate of side effects depends on the method of inserting the CVC and the skill of the operator. Previous method approached the IJV using the anatomy ladmark with the blind Seldinger technique, recently, as the use of ultrasound has become more common.

Ultra sound guided CVC insertion tecnique reduce the incidence of side effect. However, there are still major complications exist because less experiance operator inserts needle too deep without caution and only depends on the image of sonography.

Currently, the length of the needle commonly used in the CVC catheter set is 7 cm. In general, the depth from the skin to the IJV is within 1.5cm on either the right or the left, and under the premise that the needle insertion angle is 45 degrees, the distance from the skin to the IJV is within 2cm. Based on this, in previous studies, it was announced that the length of the needle required for IJV access was less than 4 cm.

The purpose of this study is to study the usefulness and safety of the method of sono-guided CVC catheter insertion by fixing the needle at a position 4 cm from the needle tip by placing the suture wing (18G, single catheter set).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who need CVC catheter for operation

Exclusion Criteria:

* Obesity (BMI > 35)
* wound or infection exist at the puncture site
* History of long term catheter placment in the IJV
* Abnormally small size or deformity of the IJV
* Past history of difiiculty in CVC catheterization

  * If the IJV is located at a depth of 3cm or more from theskin on ultrasound evaluation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-27 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The difficulty of catheterization | through study completion, an average of 10 minutes
  It would be evaluated by the operator who performed the catheterization. The severity of difficulty would be determined by total sum of the following scores.
  1. needle tip visibility with sono: good (0), not good (1), bad(2)
  2. blood aspiration was during needle withdrawal :1
  3. Number of attempt :1 ,2, 3
  Total score would be ranged from 0 to 6